CLINICAL TRIAL: NCT01561222
Title: Effect of Vitamin D Supplement on Osteoprotegin Expression and Disease Progression in Patients With Chronic Kidney Disease Stage 1 and 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taixing People's Hospital (Other)
Responsible Party: Principal Investigator, Xu Zhang, Zhang Xu, Taixing People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: zhangxu2012
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Kidney Disease Stage 1; Chronic Kidney Disease Stage 2
Keywords: calcitrol; Bone mineral density; Osteoprotegin; Vascular calcification
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vascular Calcification | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Calcitriol (Experimental)
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol — 0.25 ug per day for one year
  Other Names: Rocaltrol
  Arms: Calcitriol
Drug: placebo — one pill per day
  Arms: placebo

SUMMARY:
Vitamin D Supplement in patients with CKD stage 1 and 2 may change osteoprotegin expression so as to produce beneficial effects of cardiovascular、bone metabolism and CKD progression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CKD stage 1 and 2
* Age >18 years
* Ability to provide informed consent

Exclusion Criteria:

* On vitamin D in past 4 weeks
* Plans to relocate out of Taixing City in the next one year
* Serum phosphate >5.5 mg/dl in past 3 months
* Serum calcium >10.0 mg/dl in past 3 months
* Cancer
* Transplanted organ
* Rapidly deteriorating kidney function with the expectation for initiation of dialysis in less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Osteoprotegin level | one year
  To assess the effect of vitamin D supplementation on osteoprotegin level in CKD patients

SECONDARY OUTCOMES:
Bone mineral density | one year
  To assess the effect of vitamin D supplementation on bone mineral density in patients with CKD stage 1 and 2
vascular calcification score | one year
  To assess the effect of vitamin D supplementation on vascular calcification score through performing lateral abdominal radiography or CT-based techniques in patients with CKD stage 1 and 2

CONTACTS AND LOCATIONS:
Locations (1):
- Taixing People's Hospital, Taishing, Jiangsu, China